CLINICAL TRIAL: NCT07342231
Title: FAP-1 Study: FAPi PET in Pancreatic Ductal Adenocarcinoma: A Prospective, Exploratory Study
Brief Title: FAPi PET in Pancreatic Ductal Adenocarcinoma
Acronym: FAP-1
Status: Recruiting | Type: Observational
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Ameya Puranik, Professor, Tata Memorial Hospital
Other Study IDs: TMCIEC4238; TRAC/0324/4238/001 (Other Grant/Funding Number: DAE CTC)
Record Dates: First submitted 2025-11-19; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Cancer; Adenocarcinoma Pancreas
Keywords: Fibroblast activation protein; PETCT; FAPi
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Arm 1: Patients who have been diagnosed with pancreatic ductal adenocarcinoma will undergo Ga-: Patients with pancreatic ductal adenocarcinoma who undergo standard work-up with histopathology and conventional imaging will be referred for Ga-68 FAPi PET/CT
  Interventions: Diagnostic Test: Ga-68 FAPi PET/CT
- Study Arm 2: Treated patients with pancreatic ductal adenocarcinoma showing rising tumor markers (CA: Patients who undergo surgery or upfront chemotherapy and subsequently have rising tumor marker levels
  Interventions: Diagnostic Test: Ga-68 FAPi PET/CT

INTERVENTIONS:
Diagnostic Test: Ga-68 FAPi PET/CT — Ga-68 FAPi PET/CT is a whole body scan to assess the FAP receptor expression in patients with pancreatic ductal adenocarcinoma
  Other Names: FAPi PET

SUMMARY:
Pancreatic adenocarcinoma commonly referred to as pancreatic cancer is a cancer which is known to involve the pancreas and the surrounding structures like blood vessels, which makes it an aggressive cancer. Treatment of the cancer is decided by how much the disease has spread. It has been understood from recent studies that there are some components of the tumor which are not detected by standard CT scan. The tissue in the tumor microenvironment leads to further spread of tumor. The tissue which is seen near the tumor has many attachments on the surface which are currently being studied. One of the most common attachments is Fibroblast activation protein (FAP), which is seen on the surface of tumor tissue. A radioactive tracer Gallium-68 is attached to a small protein known as 'peptide' named 'FAP inhibitor (FAPi)' which shall bind to FAP. Then a PET scan will be performed which shall help in understanding how much of the tissue is seen on the scan in addition to the pancreatic tumor. The investigators shall assess whether the radiotracer (Gallium-68 labeled FAPi) binds to other sites like liver or other organs where the cancer is likely to spread. From the study, the investigators shall study whether the new scanning technique is beneficial as compared to the standard CT scanning. Hence, the investigators would perform Gallium-68-labeled FAPi PET scan in addition to the standard CT scan and compare the results.

ELIGIBILITY:
Inclusion Criteria:

* Any gender with age more than 18 years
* Patients with biopsy-proven pancreatic ductal adenocarcinoma
* Patient willing to participate in study

Exclusion Criteria:

* Patient with concurrent malignancy
* Pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with biopsy proven pancreatic ductal adenocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-01-04 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Imaging validation of Ga-68 FAPi PET/CT | 6 and 12 months
  To calculate sensitivity, specificity, positive predictive value and negative predictive value of quantitative and semi-quantitative parameters on FAPi PET

CONTACTS AND LOCATIONS:
Overall Officials: Ameya Puranik, DNB, Principal Investigator — Tata Memorial Hospital, Mumbai
Locations (1):
- Tata Memorial Hospital, Mumbai, India, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No
It is against the recommendations of institutional ethics committee

REFERENCES:
- [Background] Yuan H, Liu E, Zhang G, Lai C, Zhang Q, Shang Y, Cheng Z, Jiang L. Diagnostic efficacy of [68Ga]Ga-DOTA-GPFAPI-04 in patients with solid tumors in a head-to-head comparison with [18F]F-FDG: results from a prospective clinical study. Eur J Nucl Med Mol Imaging. 2024 Sep;51(11):3360-3372. doi: 10.1007/s00259-024-06756-0. Epub 2024 May 10. PMID 38727829

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT07342231/Prot_SAP_000.pdf